CLINICAL TRIAL: NCT06413719
Title: Assessing the Effects of Chiropractic Care in Children With Parent-reported Sensory Processing Disorder: a Feasibility Study
Brief Title: Assessing the Effects of Chiropractic Care in Children With Parent-reported Sensory Processing Disorder
Acronym: SPD
Status: Withdrawn | Type: Observational
Why Stopped: Study designed changed to observational study
Sponsor: Life University (Other)
Responsible Party: Sponsor
Other Study IDs: I-0030
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sensation Disorders
Keywords: Pediatrics; sensation disorders; autonomic nervous system; HRV; heart rate variability
MeSH Terms: conditions — Sensation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Intervention: Children with probable or definite sensory processing challenges per the SSP-1

SUMMARY:
This trial's main aims are to investigate the feasibility of implementing our novel assessment battery in tandem with normal and customary chiropractic care in a practice-based setting using a pediatric population with parent-reported SPD. More specifically, our primary endpoints are 1) recruitment rate, 2) tolerability, 3) adherence, 4) retention, 5) efficiency, and 6) data quality.

DETAILED DESCRIPTION:
The total estimated time requirement for this study is ~60 minutes.

Up to 20 children (ages 5-12) will be recruited in a maximum 3-month enrollment period. The total estimated time requirement for the parent and child is ~1 hour excluding the normal and customary chiropractic care. Per the clinic's normal and customary procedures, a welcome email is sent to each parent who schedules their child for a chiropractic exam at Premier Wellness Care (PWC) chiropractic (Crystal Lake, IL). An addendum will be added to this email briefly introducing the study along with a HIPAA compliant Jotform link to an online screening survey which incorporates the 38-item short sensory profile v1 (SSP-1). Those who complete the online screen and meet the eligibility criteria described below will be notified when they arrive at PWC for their initial exam & offered the opportunity to participate in the study.

Informed consent (IC) and assent (IA) will be collected in a private room within PWC. A PWC staff member (TM) will sit down with each parent & child to review the IC & IA forms and answer any queries. To be enrolled, the parent must sign the IC and the child must acknowledge their willingness to participate verbally (e.g., "yes I would like to do the study") and/or physically (e.g., nod their head & give a 'thumbs up'). It will be made clear to all parents & children that they may decline participation without penalty and declining participation will in no way impact the child's access to normal and customary chiropractic care.

Children will be asked to stand up straight on a scale so the investigators can measure their heights and weights. They will then be asked to sit in a comfortable chair, shown a visual analog scale (VAS), and asked to rate their pain level on a scale from 0 ("no pain") to 10 ("worst pain possible").

To track autonomic nervous system (ANS) activity, children will be asked to place their hand on the class II FDA registered neuroPULSE scanner (CLA Inc., Toronto, ON, Canada) and put their index, middle, & ring fingers onto the sensors. To track sweat gland (i.e., electrodermal, EDA) activity, a safe and unrecognizable low-voltage, high-amplitude current is passed between sensors located at the palmar-surfaces of the index and ring fingers. The pulse rate is measured via photoplethysmography (PPG) whereby blood flow-dependent changes in the quantity of emitted light passing though the fingertip are tracked via a sensor located on the palmar-surface of the middle finger. All signals will be transmitted to an iPad for viewing by the assessor via a secure Wi-Fi connection.

With their hand in the neuroPULSE, children will undergo a sensory challenge protocol (SCP). For the SCP, the kids will be fitted with noise cancelling headphones and be shown a series of pictures. Prior to initiating the SCP, the assessor will instruct the child how to perform the test. The headphones will then be paired via Bluetooth to an iPhone/iPad device & switched on. Upon presentation of the "sitting" picture, the child will be asked to sit still and quietly for ~2 minutes. Upon presentation of the "standing" picture, they will be asked to quickly stand and remain still and quiet for ~2 minutes. Upon re-presentation of the "sitting" picture, the child will be asked to quickly return to a seated position & remain still and quiet for ~2 minutes. Finally, upon presentation of the "noise" picture, the child will be asked to sit still and quietly while an auditory stimulus (1000 Hz, sine wave, 50% system volume, ~75 dB) generated via a free tone generator app (f Generator, v7.4.1) is presented to both ears through the headphones for ~2 minutes. The sound is like what someone would hear on your mobile device during an "AMBER Alert". This prolonged auditory stimulus is well below acceptable noise exposure limits and is in line with a protocol used in prior studies to test pediatric SPD populations. To help keep the children occupied during the SCP, a researcher will place an iPad directly in front of the subject & play a relaxing video (e.g., fish swimming in the ocean). When the SCP is finished, the video will be stopped, the headphones will be removed, and the child will be asked to remove his/her hand from the neuroPULSE scanner. During the child's assessment, parents will then be given an iPad & asked to complete the 38-item SSP-1.

All assessments will be repeated following 12 sessions of PWC's normal and customary chiropractic care.

ELIGIBILITY:
Inclusion Criteria:

* 5-12 years of age
* SSP-1 total score no greater than 154

Exclusion Criteria:

* Unable to perform assessments due to vision, hearing, or movement impairment (e.g., blind, deaf, confined to wheelchair)
* Unable to perform the assessments due to a preexisting condition whereby quick postural changes are contraindicated (e.g., postural orthostatic tachycardia syndrome (POTS), postural hypotension)
* Pacemaker or known heart condition that influences the electrical or mechanical function of the heart

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with probable or definite sensory processing challenges per the SSP-1
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 3 months (recruitment period)
  Average number of subjects enrolled per month
Tolerability | 4 months (data collection period)
  % of participants unable/unwilling to tolerate (i.e., complete as directed) a given assessment
Adherence | 4 months (data collection period)
  % of participants attending <80% of their chiropractic sessions within the recommended time frame
Retention | 4 months (data collection period)
  % of participants completing the trial
Efficiency | 4 months (data collection period)
  Average time to completion of each assessment section
Data quality | 6 months (study period)
  % of acquisitions unsuitable for analysis for a given assessment

CONTACTS AND LOCATIONS:
Overall Officials: Tyson Perez, DC, PhD, Principal Investigator — Life University

IPD SHARING:
Plan to Share IPD: No